CLINICAL TRIAL: NCT00980135
Title: An Investigator-blind, Randomized, Monocentre, 3-arm, Active Controlled Pilot Trial to Explore the Efficacy and Safety of a New Topical Medical Device in Patients With Mild Atopic Dermatitis in an Intra-individual Comparison With a Standard Therapy (1% Hydrocortisone Cream) and Untreated Skin.
Brief Title: Sinecort Pilot Efficacy Study
Acronym: Sinecort Pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13932; 2008-008136-82 (EudraCT Number)
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Atopic Dermatitis
Keywords: Sinecort; Hydrocortison; Mild atopic dermatitis; Efficacy, safety
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Device: Sinecort cream
- Arm 2 (Experimental)
  Interventions: Drug: Hydrocortison cream
- Arm 3 (Other)
  Interventions: Other: Untreated skin

INTERVENTIONS:
Device: Sinecort cream — Application over 29 days
  Arms: Arm 1
Drug: Hydrocortison cream — Application over 29 days
  Arms: Arm 2
Other: Untreated skin
  Arms: Arm 3

SUMMARY:
The study shall prove whether treatment of atopic dermatitis is equally effective with Sinecort cream as compared to standard therapy (Hydrocortisone cream).

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasians aged between 18 and 65 years
* Patients with mild AD presenting a scoring AD (SCORAD) rating between 3-25
* Skin type I - IV according to Fitzpatrick
* Acute AD symptoms on each assessment areas (local SCORAD >/=3 and <= 12)
* Acute symptom of pruritus at Baseline

Exclusion Criteria:

* Any other skin disease at the test area that would interfere the clinical assessment in the opinion of the investigator
* Moles, tattoos, strong pigmentation, or scars at the test area that would interfere the clinical assessment
* Regular intake of antiphlogistic drugs (for example, NSAIDs)
* Any condition or treatment which might influence the trial (e.g. any treatment with topical antibiotics, antifungals, or corticoids) within 14 days prior to screening as well as during the trial (exception: topical treatment of AD lesions other than the test areas (for example, face) with low potency steroids restricted to small areas)
* UV-therapy or the use of solarium within 30 days before screening as well as during the trial
* Any alternative treatment of AD (e.g. acupuncture, kinesiology, and homoeopathy) within 30 days before screening as well as during the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Efficacy rate versus comparator and untreated skin | After 29 days of twice daily applications
Local side effects on the skin | 29 days

SECONDARY OUTCOMES:
Local SCORAD as clinical assessment by means of the intensity items of the SCORAD index) at Visit 2 through Visit 6 | after 29 days
Transepidermal water loss (TEWL) as a measure for skin barrier function at Visit 2 through Visit 6 | after 29 days
Skin hydration by means of corneometry at visit 2 through visit 6 | after 29 days
Erythema by means of chromametry at Visit 2 through Visit 6 | after 29 days
Intensity of pruritus at each day of the dosing period (day 1- day 29) as reported in the patients diary and at Visit 2 through Vist 6 by means of visual analogue scale (VAS) | after 29 days
Incidence and severity of Adverse Event | visit 2 (start of dosing period) till 6 weeks after end of treatment
Vital signs | visit1 and 6 weeks after end of treatment
Local side effects | visit 2 (start of dosing period) till 6 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Münster, North Rhine-Westphalia, Germany